CLINICAL TRIAL: NCT03489148
Title: Implications of Tamarkoz® on Reducing Stress and Heart Rate, and Increasing Positive Emotions, Spirituality
Brief Title: Implications of Tamarkoz® on Stress, Emotion, Spirituality and Heart Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5150225
Record Dates: First submitted 2018-03-04; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Stress
Keywords: Stress; Relaxation; Health promotion

STUDY DESIGN:
Intervention Model Description: Participants were recruited from the University of California, Berkeley for an 18-week quasi-experimental study with pretest-posttest and follow-up in three groups. Assessments were conducted with blood pressure, heart rate, the 10-item perceived stress scale, the 38-item dispositional positive emotions scale, and the 16-item daily spiritual experiences scale in a Tamarkoz® group, a wait-list control, and a third group utilizing the campus health center's stress management resources. Blood pressure and heart rate measurements were taken by the researcher using a validated home monitoring device. Additionally, all participants provided 3 diurnal saliva samples to determine changes in salivary immunoglobulin A and salivary cortisol. All data were collection was through non-evasive procedures and were assessed at baseline, end of the school semester (12 weeks) and 18 weeks.
Who Masked: Care Provider
Masking Description: The Tamarkoz® class instructor was not informed about which of her students from the class was participating in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tamarkoz® (Experimental): A Sufi method to focus, called Tamarkoz®. Participants had met in class twice a week for two and a half hours total for three months. One day of the week, they met for theoretical teachings of Sufism, and for the second day in the week they met with a Tamarkoz® instructor to learn meditation techniques.
  Interventions: Behavioral: Tamarkoz®
- Stress Management Resources (Active Comparator): The self-care stress management group used the campus resources such as counseling, health-coaching, health and wellness groups, use of an automated massage chair, and online reading materials for stress management as needed for themselves.
  Interventions: Behavioral: Stress management resources
- Waitlist (No Intervention): The waitlist control group did not receive Tamarkoz® and did not use the stress management resources on campus for the duration of the study.

INTERVENTIONS:
Behavioral: Tamarkoz® — Tamarkoz® techniques includes six key elements: clearing the mind, breathing exercises, Movazeneh® (movement and balance exercises), deep relaxation, and visualization.
  Arms: Tamarkoz®
Behavioral: Stress management resources — Use of the campus health center's stress management resources such as counseling, health-coaching, health and wellness groups, use of an automated massage chair, pet-an-animal a week, and online reading material about self-care for stress management.
  Arms: Stress Management Resources

SUMMARY:
Depression, anxiety, hopelessness, poor sleep quality, somatic pain, high risk of substance abuse, and suicide ideation are positively correlated with perceived stress. Spirituality and positive emotions have profound, positive impacts on health and reduce perceived stress. The current study is an exploration of Tamarkoz®, a Sufi practice that is a method to concentrate, as a pathway by which spirituality and positive emotions effect perceived stress. Tamarkoz® incorporates physical, emotional, and spiritual aspects of an individual. In its current form, it includes Movazaneh® which is movement balancing developed by the Sufi Master, Professor Nader Angha. Movazaneh® movements direct concentration of the mind to a state of collectiveness and activates electromagnetic centers in the body, which are said to develop spirituality in an individual. A national survey of college students indicated that over 80% have interest in spiritual development.

Participants were recruited from the University of California, Berkeley for an 18-week quasi-experimental study with pretest-posttest and follow-up in three groups. Assessments were conducted with blood pressure, heart rate, the 10-item perceived stress scale, the 38-item dispositional positive emotions scale, and the 16-item daily spiritual experiences scale in a Tamarkoz® group, a wait-list control, and a third group utilizing the campus health center's stress management resources. Blood pressure and heart rate measurements were taken by the researcher using a validated home monitoring device. Additionally, all participants provided 3 diurnal saliva samples to determine changes in salivary immunoglobulin A and salivary cortisol. All data were collection was through non-evasive procedures and were assessed at baseline, end of the school semester (12 weeks) and 18 weeks.

Participants, diverse university students, had no prior exposure to Tamarkoz®.

DETAILED DESCRIPTION:
This study is quasi-experimental, waitlist control group design with pretest-posttest. It consisted of three groups: (a) the intervention group who learned Tamarkoz® Sufi meditation practices, (b) a second group of students who utilized self-care stress management resources at the Tang University Health Services Center, and (c) a third group who was the waitlist control group who did not receive Tamarkoz® and did not use the stress management resources at the Tang Center for the duration of the study.

The design is represented in the following diagram. NR O(a) XT O(b) O(d) NR O(d) XS O(e) O(g) NR O(g) O(h) O(i)

XT represents twelve weeks of Tamarkoz® training and XS represents twelve weeks of Tang Center stress management techniques. Each O represents one of three measurements in each group: (a) at baseline, (b) 12 weeks later, immediately after the intervention ends, and (c) six weeks post-intervention. The intervention group met twice a week for two and a half hours total for three months. One day of the week, they met for theoretical teachings of Sufism, and for the second day in the week they met to learn Tamarkoz® techniques. The self-care stress management group used the campus resources for stress management as needed for themselves.

ELIGIBILITY:
Inclusion Criteria:

* University of California, Berkeley students between the ages of 18-30 years

Exclusion Criteria:

* work third shifts
* diabetes
* post-traumatic stress disorder
* liver disease
* autoimmune diseases
* severe depression that resists treatment or impacts ability to function
* schizophrenia

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2016-02-04 (Actual); Study Completion 2016-02-04 (Actual)

PRIMARY OUTCOMES:
Perceived stress scale | Change between baseline and 18 weeks
  The scale measures the degree to which one perceives situations in one's life as stressful on a Likert Scale of 0 to 4 with 0 indicating never, and 4 indicating very often. Higher scores indicate higher levels of perceived stress.

SECONDARY OUTCOMES:
Salivary Immunoglobulin A (SIgA) in Saliva | Change between baseline and 18 weeks
  Analysis of saliva drool analysis of salivary immunoglobbulin A immune cell. Lab will analyze the saliva. Normal levels of SIgA have not been determine.

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Bahadorani, DrPH, Principal Investigator — Loma Linda University; Jerry W Lee, PhD, Study Chair — Loma Linda University
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 6 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Largo-Wight E, Peterson PM, Chen WW. Perceived problem solving, stress, and health among college students. Am J Health Behav. 2005 Jul-Aug;29(4):360-70. doi: 10.5993/ajhb.29.4.8. PMID 16006233
- [Background] Bayram N, Bilgel N. The prevalence and socio-demographic correlations of depression, anxiety and stress among a group of university students. Soc Psychiatry Psychiatr Epidemiol. 2008 Aug;43(8):667-72. doi: 10.1007/s00127-008-0345-x. Epub 2008 Apr 8. PMID 18398558
- [Background] Devos, C., Boudrenghien, G., Van der Linden, N., Azzi, A., Frenay, M., Galand, B., & Klein, O. Doctoral students' experiences leading to completion or attrition: A matter of sense, progress and distress. European Journal of Psychology of Education: 1-17, 2016. doi:10.1007/s10212-016-0290-0
- [Background] Romans, J. S. C., White, J. K., Harrist, R. S., Boswell, D. L., Sims, W. D., & Murn, L. T. Predicting attrition from counseling in a university counseling center sample using the Outcome Questionnaire-45.2. Internet Journal of Mental Health, 7(1), 1-8, 2011.
- [Background] Lund HG, Reider BD, Whiting AB, Prichard JR. Sleep patterns and predictors of disturbed sleep in a large population of college students. J Adolesc Health. 2010 Feb;46(2):124-32. doi: 10.1016/j.jadohealth.2009.06.016. Epub 2009 Aug 3. PMID 20113918
- [Background] Kennedy C, Kassab O, Gilkey D, Linnel S, Morris D. Psychosocial factors and low back pain among college students. J Am Coll Health. 2008 Sep-Oct;57(2):191-5. doi: 10.3200/JACH.57.2.191-196. PMID 18809536
- [Background] Dixon, W. A., Rumford, K. G., Heppner, P. P., & Lips, B. J. Use of different sources of stress to predict hopelessness and suicide ideation in a college population. Journal of Counseling Psychology, 39(3), 342-349, 1992. doi:10.1037/0022-0167.39.3.342
- [Background] Oman D, Shapiro SL, Thoresen CE, Plante TG, Flinders T. Meditation lowers stress and supports forgiveness among college students: a randomized controlled trial. J Am Coll Health. 2008 Mar-Apr;56(5):569-78. doi: 10.3200/JACH.56.5.569-578. PMID 18400671
- [Background] Mahmoud JS, Staten R, Hall LA, Lennie TA. The relationship among young adult college students' depression, anxiety, stress, demographics, life satisfaction, and coping styles. Issues Ment Health Nurs. 2012 Mar;33(3):149-56. doi: 10.3109/01612840.2011.632708. PMID 22364426
- [Background] O'Leary A. Stress, emotion, and human immune function. Psychol Bull. 1990 Nov;108(3):363-82. doi: 10.1037/0033-2909.108.3.363. PMID 2270233
- [Background] Herman L, Shtayermman O, Aksnes B, Anzalone M, Cormerais A, Liodice C. The use of prescription stimulants to enhance academic performance among college students in health care programs. J Physician Assist Educ. 2011;22(4):15-22. doi: 10.1097/01367895-201122040-00003. PMID 22308929
- [Background] Sawatzky RG, Ratner PA, Richardson CG, Washburn C, Sudmant W, Mirwaldt P. Stress and depression in students: the mediating role of stress management self-efficacy. Nurs Res. 2012 Jan-Feb;61(1):13-21. doi: 10.1097/NNR.0b013e31823b1440. PMID 22166906
- [Background] Taub, D. J., & Thompson, J. College Student Suicide. New Directions for Student Services, 2013(141), 5-14, 2013. doi:10.1002/ss.20036
- [Background] Adams DR, Meyers SA, Beidas RS. The relationship between financial strain, perceived stress, psychological symptoms, and academic and social integration in undergraduate students. J Am Coll Health. 2016 Jul;64(5):362-70. doi: 10.1080/07448481.2016.1154559. Epub 2016 Mar 4. PMID 26943354
- [Background] DeRoma, V. M., Leach, J. B., & Leverett, J. P. The relationship between depression and college academic performance. College Student Journal, 43(2), 325-334, 2009
- [Background] Oman D, Hedberg J, Thoresen CE. Passage meditation reduces perceived stress in health professionals: a randomized, controlled trial. J Consult Clin Psychol. 2006 Aug;74(4):714-9. doi: 10.1037/0022-006X.74.4.714. PMID 16881779
- [Background] Struthers, C. W., Perry, R. P., & Menec, V. H. An Examination of the Relationship Among Academic Stress, Coping, Motivation, and Performance in College. Research in Higher Education, 41(5), 581-592, 2000. doi:10.1023/a:1007094931292
- [Background] Aselton P. Sources of stress and coping in American college students who have been diagnosed with depression. J Child Adolesc Psychiatr Nurs. 2012 Aug;25(3):119-23. doi: 10.1111/j.1744-6171.2012.00341.x. Epub 2012 Jul 2. PMID 22830509
- [Background] Dusselier L, Dunn B, Wang Y, Shelley MC 2nd, Whalen DF. Personal, health, academic, and environmental predictors of stress for residence hall students. J Am Coll Health. 2005 Jul-Aug;54(1):15-24. doi: 10.3200/JACH.54.1.15-24. PMID 16050324
- [Background] Kitzrow, M. A. The mental health needs of today's college students: Challenges and recommendations. Journal of Student Affairs Research and Practice, 41(1), 165-179, 2003.
- [Background] Watkins, D. C., Hunt, J. B., & Eisenberg, D. Increased demand for mental health services on college campuses: Perspectives from administrators. Qualitative Social Work, 11(3), 319-337, 2012.
- [Background] Burns, J. L., Lee, R. M., & Brown, L. J. The Effect of Meditation on Self-Reported Measures of Stress, Anxiety, Depression, and Perfectionism in a College Population. Journal of College Student Psychotherapy, 25(2), 132-144, 2011. doi:10.1080/87568225.2011.556947
- [Background] Ratanasiripong, P., Sverduk, K., Hayashino, D., & Prince, J. Setting up the next generation biofeedback program for stress and anxiety management for college students: a simple and cost-effective approach. College Student Journal, 44(1), 97, 2010.
- [Background] Paul G, Elam B, Verhulst SJ. A longitudinal study of students' perceptions of using deep breathing meditation to reduce testing stresses. Teach Learn Med. 2007 Summer;19(3):287-92. doi: 10.1080/10401330701366754. PMID 17594225
- [Background] Kirk U, Downar J, Montague PR. Interoception drives increased rational decision-making in meditators playing the ultimatum game. Front Neurosci. 2011 Apr 18;5:49. doi: 10.3389/fnins.2011.00049. eCollection 2011. PMID 21559066
- [Background] Ramsburg, J., & Youmans, R. Meditation in the Higher-Education Classroom: Meditation Training Improves Student Knowledge Retention during Lectures. Mindfulness, 1-11, 2013. doi:10.1007/s12671-013-0199-5
- [Background] So, K.-T., & Orme-Johnson, D. W. Three randomized experiments on the longitudinal effects of the Transcendental Meditation technique on cognition. Intelligence, 29(5), 419-440, 2001. doi:http://dx.doi.org/10.1016/S0160-2896(01)00070-8
- [Background] Wachholtz AB, Pargament KI. Is spirituality a critical ingredient of meditation? Comparing the effects of spiritual meditation, secular meditation, and relaxation on spiritual, psychological, cardiac, and pain outcomes. J Behav Med. 2005 Aug;28(4):369-84. doi: 10.1007/s10865-005-9008-5. PMID 16049627
- [Background] Miller WR, Thoresen CE. Spirituality, religion, and health. An emerging research field. Am Psychol. 2003 Jan;58(1):24-35. doi: 10.1037/0003-066x.58.1.24. PMID 12674816
- [Background] Angha, N. (2002). Theory
- [Background] Angha, S. A. N. (2000). Expansion and Contraction Within Being (Dahm). Riverside, California: M.T.O. Shahmaghsoudi Printing and Publication Center.
- [Background] Dein, S. Religion, spirituality and depression: Implications for research and treatment. Primary Care and Community Psychiatry, 11, 67 - 72, 2006.
- [Background] Carmody J, Reed G, Kristeller J, Merriam P. Mindfulness, spirituality, and health-related symptoms. J Psychosom Res. 2008 Apr;64(4):393-403. doi: 10.1016/j.jpsychores.2007.06.015. Epub 2008 Mar 4. PMID 18374738
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Shiota, M., Dacher, K., & Oliver, J. Positive emotion dispositions differentially associated with Big Five personality and attachment style. The Journal of Positive Psychology, 1(2), 61-71, 2006.
- [Background] Underwood. The Daily Spiritual Experience Scale: Overview and Results. Religions, 2(1), 29-50, 2011.
- [Background] Cohen, S., & Janicki-Deverts, D. Who's stressed? Distributions of psychological stress in the United States in probability samples from 1983, 2006, and 2009. Journal of Applied Social Psychology, 42(6), 1320-1334, 2012.
- [Background] Stellar JE, John-Henderson N, Anderson CL, Gordon AM, McNeil GD, Keltner D. Positive affect and markers of inflammation: discrete positive emotions predict lower levels of inflammatory cytokines. Emotion. 2015 Apr;15(2):129-33. doi: 10.1037/emo0000033. Epub 2015 Jan 19. PMID 25603133
- [Background] Stewart-Brown S, Evans J, Patterson J, Petersen S, Doll H, Balding J, Regis D. The health of students in institutes of higher education: an important and neglected public health problem? J Public Health Med. 2000 Dec;22(4):492-9. doi: 10.1093/pubmed/22.4.492. PMID 11192277
- [Background] Fredrickson BL. What Good Are Positive Emotions? Rev Gen Psychol. 1998 Sep;2(3):300-319. doi: 10.1037/1089-2680.2.3.300. PMID 21850154
- [Background] Fredrickson BL. The role of positive emotions in positive psychology. The broaden-and-build theory of positive emotions. Am Psychol. 2001 Mar;56(3):218-26. doi: 10.1037//0003-066x.56.3.218. PMID 11315248
- [Background] Tugade MM, Fredrickson BL. Resilient individuals use positive emotions to bounce back from negative emotional experiences. J Pers Soc Psychol. 2004 Feb;86(2):320-33. doi: 10.1037/0022-3514.86.2.320. PMID 14769087
- [Background] Kim, Y., & Seidlitz, L. Spirituality moderates the effect of stress on emotional and physical adjustment. Personality & Individual Differences, 32(8), 1377, 2002.
- [Background] Powers, D. V., Cramer, R. J., & Grubka, J. M. Spirituality, life stress, and affective well-being. Journal of Psychology and Theology, 35(3), 235, 2007.
- [Background] Chang BH, Casey A, Dusek JA, Benson H. Relaxation response and spirituality: Pathways to improve psychological outcomes in cardiac rehabilitation. J Psychosom Res. 2010 Aug;69(2):93-100. doi: 10.1016/j.jpsychores.2010.01.007. Epub 2010 Mar 1. PMID 20624507
- [Background] Hill PC, Pargament KI. Advances in the conceptualization and measurement of religion and spirituality. Implications for physical and mental health research. Am Psychol. 2003 Jan;58(1):64-74. doi: 10.1037/0003-066x.58.1.64. PMID 12674819
- [Background] Tuck I, Alleyne R, Thinganjana W. Spirituality and stress management in healthy adults. J Holist Nurs. 2006 Dec;24(4):245-53; discussion 254-5. doi: 10.1177/0898010106289842. PMID 17098877
- [Background] Keefe FJ, Affleck G, Lefebvre J, Underwood L, Caldwell DS, Drew J, Egert J, Gibson J, Pargament K. Living with rheumatoid arthritis: the role of daily spirituality and daily religious and spiritual coping. J Pain. 2001 Apr;2(2):101-10. doi: 10.1054/jpai.2001.19296. PMID 14622831
- [Derived] Bahadorani N, Lee JW, Martin LR. Implications of Tamarkoz on stress, emotion, spirituality and heart rate. Sci Rep. 2021 Jul 8;11(1):14142. doi: 10.1038/s41598-021-93470-8. PMID 34238979
- See also: M.T.O.®. (2016). Tamarkoz® — http://tamarkoz.org
- See also: Higher Education Research Institute. (2007). The spiritual life of college students: A national study of college students' search for meaning and purpose — http://spirituality.ucla.edu/docs/reports/Spiritual_Life_College_Students_Full_Report.pdf
- See also: Smith, T. W., Hout, M., & Marsden, P. V. (2013). General Social Survey, 1972-2012 — http://doi.org/10.3886/ICPSR34802.v1